CLINICAL TRIAL: NCT06004804
Title: Evaluating Group-Based Psychological Treatments Over Home Video Teleconference for Older Veterans With Chronic Pain
Brief Title: Group-Based Psychological Treatments Over Video Conference for Older Veterans With Chronic Pain
Acronym: GPTVTCOVCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 21-207; I01HX003494-01A2 (NIH)
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Chronic pain; Psychological intervention; Musculoskeletal disease; Telehealth
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Diseases | interventions — Mindfulness; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Three-Group Parallel Comparison Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study will rely on a blinded outcomes assessor who will be blind to condition assignment. Investigators will be blind to outcomes until the conclusion of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Emotional Awareness and Expression Therapy (Experimental): Seeks to reduce physical (e.g., pain) and emotional (e.g., depression, anxiety) symptoms by helping individuals become aware of their emotions, express them, and resolve emotional conflicts. It will use techniques such as writing about stress, role playing how to handle difficult relationships, recognizing and expressing anger and other feelings, and being more open with others.
  Interventions: Behavioral: Emotional Awareness and Expression Therapy
- Mindfulness Meditation (Experimental): Seeks to help individuals achieve present moment awareness, self-compassion, and acceptance of chronic pain. It will use techniques such as the body scan, grounding, mindful breathing, mindful walking, loving kindness, and compassionate breathing.
  Interventions: Behavioral: Mindfulness Meditation
- Cognitive Behavioral Therapy (Active Comparator): Seeks to help individuals function better and improve symptoms by teaching various cognitive and behavioral skills to manage symptoms. It will use techniques such as relaxation training, engaging in pleasant activities, pacing yourself, and changing unhelpful ways of thinking.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy — Seeks to reduce physical (e.g., pain) and emotional (e.g., depression, anxiety) symptoms by helping individuals become aware of their emotions, express them, and resolve emotional conflicts. It will use techniques such as writing about stress, role playing how to handle difficult relationships, recognizing and expressing anger and other feelings, and being more open with others.
  Other Names: EAET
  Arms: Emotional Awareness and Expression Therapy
Behavioral: Mindfulness Meditation — Seeks to help individuals achieve present moment awareness, self-compassion, and acceptance of chronic pain. It will use techniques such as the body scan, grounding, mindful breathing, mindful walking, loving kindness, and compassionate breathing.
  Other Names: MM
  Arms: Mindfulness Meditation
Behavioral: Cognitive Behavioral Therapy — Seeks to help individuals function better and improve symptoms by teaching various cognitive and behavioral skills to manage symptoms. It will use techniques such as relaxation training, engaging in pleasant activities, pacing yourself, and changing unhelpful ways of thinking.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This study is being performed to compare the effects of three types of group-based psychological treatments delivered over video telehealth for chronic musculoskeletal pain in older U.S. military Veterans. The three types of psychological treatments are: Cognitive-Behavioral Therapy (CBT), Emotional Awareness and Expression Therapy (EAET), and Mindfulness Meditation (MM). In addition, the investigators will evaluate which patients respond best to each treatment and how each treatment works.

The investigators are performing the study because chronic pain is a big problem among Veterans. Older Veterans are the focus because they have the highest rates of chronic pain, perhaps as high has 80%. The investigators are looking at psychological treatments because they are less risky than medications or procedures for older Veterans. Telehealth is an important aspect of the proposal, as delivery over telehealth could improve access to treatments. CBT is endorsed nationally by VA, but no standardized MM is available through VA, and only a few VA sites use EAET, which is a newer treatment focusing on how stress and emotions affect pain. The project aims to evaluate a standardized form of MM and the newer treatment, EAET, compared to the standard CBT used widely in VA.

DETAILED DESCRIPTION:
The overarching goal of the proposed research is to learn how to optimize group-based psychological treatments for chronic pain delivered over video telehealth to the homes of older Veterans. Chronic pain is a critical healthcare challenge for VA, because the condition affects 50% of Veterans and is notoriously difficult to treat. Older Veterans are affected with chronic pain even more commonly and severely than younger Veterans, and older Veterans are more susceptible to side effects from pain medications and invasive procedures. Psychological chronic pain treatments do not usually have severe side effects, but tend to produce only modest benefits. To increase the effectiveness of psychological treatments, VA experts have recommended testing standardized treatments with larger and more durable benefits, testing group and video telehealth delivered treatments to improve access, identifying mechanisms of response so that the most powerful mechanisms may be targeted, and determining what Veteran characteristics may predict response to the various treatment options. The proposed randomized clinical trial will address all the recommendation of VA experts. First, the project will evaluate the effects of standardized formats of Mindfulness Meditation (MM) and Emotional Awareness and Expression Therapy (EAET) compared to the VA standard psychological chronic pain treatment, Cognitive Behavioral Therapy (CBT). Many Veterans are interested in MM, but a standardized protocol so far has not been established. EAET is a newer treatment that addresses painful stress and emotions to reduce or eliminate chronic pain. These two approaches are hypothesized to have larger benefits than CBT. Second, the project will deliver all treatments in groups and over video telehealth to the homes of Veterans to enhance access. Third, the project will test shared and specific (unique) mechanisms of response for each treatment. Fourth, the project will evaluate a set of demographic and clinical characteristics (e.g., trauma history) to see whether Veterans with certain characteristics are more likely to respond to one treatment or another. The Investigators plan to enroll up to 216 multi-ethnic/multi-racial older Veterans (age 60-95 years) with chronic musculoskeletal pain at VA Greater Los Angeles Healthcare System and VA Connecticut Healthcare System.

ELIGIBILITY:
Inclusion Criteria:

Eligible individuals are

* Veterans;
* age 60-95 years;
* have at least 3 months of musculoskeletal pain, including the following conditions: back, neck, leg, or pelvic pain; temporomandibular joint disorders; fibromyalgia; tension headaches; or any combination of these disorders; and
* have an average daily pain intensity of at least 4 on a 0 to 10 scale.

Exclusion Criteria:

* pain conditions likely to respond pharmacologic or surgical treatment only when they are the primary or sole complaint: hip or knee osteoarthritis, leg pain greater than back pain (to exclude radiculopathy), electromyography-confirmed "tunnel" syndromes (e.g., carpal tunnel syndrome), gout, neuralgias, migraine, and cluster headaches;
* non-musculoskeletal pain conditions: autoimmune disease that typically generates pain (e.g., rheumatoid arthritis), cancer pain, sickle cell disease, burn pain, infection associated with pain, and cauda equina syndrome; and
* these conditions or circumstances: severe psychiatric disorder such as schizophrenia or bipolar I disorder not controlled with medications, active suicide or violence risk, active severe alcohol or substance use disorder, substantial cognitive impairment or dementia (assessed using telephone Mini-Mental State Examination (tMMSE) score <19), previously completed EAET, CBT-CP, or MM/MBSR, currently enrolled in another psychological pain treatment, currently in pain-related litigation or applying for pain-related compensation or compensation increase, unable to fluently read or converse in English, no home internet access.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory: Mean Pain Severity | Change from baseline to 8 weeks
  Average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10.
Brief Pain Inventory: Mean Pain Severity | Change from baseline to 20 weeks
  Average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10.

SECONDARY OUTCOMES:
Brief Pain Inventory: Pain Interference | Change from baseline to 8 weeks
  Average of 7 self report items on interference of pain with daily activities over the last 7 days: general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. Each item is scored 0-10 (0 = does not interfere; 10 = completely interferes), yielding a total score between 0 and 10.
Brief Pain Inventory: Pain Interference | Change from baseline to 20 weeks
  Average of 7 self report items on interference of pain with daily activities over the last 7 days: general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. Each item is scored 0-10 (0 = does not interfere; 10 = completely interferes), yielding a total score between 0 and 10.
Patient Health Questionnaire-8 | Change from baseline to 8 weeks
  Sum of 8 self report items assessing depression and emotional distress over the last 2 weeks. Items range from 0-3 (0 = not at all; 3 = nearly every day) for a total score between 0 and 24.
Patient Health Questionnaire-8 | Change from baseline to 20 weeks
  Sum of 8 self report items assessing depression and emotional distress over the last 2 weeks. Items range from 0-3 (0 = not at all; 3 = nearly every day) for a total score between 0 and 24.
Generalized Anxiety Disorder 7-item | Change from baseline to 8 weeks
  Sum of 7 self report items assessing anxiety and worrying over the last 2 weeks. Items range from 0-3 (0 = not at all; 3 = nearly every day) for a total score between 0 and 21.
Generalized Anxiety Disorder 7-item | Change from baseline to 20 weeks
  Sum of 7 self report items assessing anxiety and worrying over the last 2 weeks. Items range from 0-3 (0 = not at all; 3 = nearly every day) for a total score between 0 and 21.
PTSD Checklist for DSM-5 | Change from baseline to 8 weeks
  Sum of 20 self report items assessing post-traumatic stress disorder symptoms over the last month. Items range from 0-4 (0 = not at all; 3 = extremely) for a total score between 0 and 80.
PTSD Checklist for DSM-5 | Change from baseline to 20 weeks
  Sum of 20 self report items assessing post-traumatic stress disorder symptoms over the last month. Items range from 0-4 (0 = not at all; 3 = extremely) for a total score between 0 and 80.
Patient's Global Impression of Change | 8 weeks
  Patient rates on a single item with a scale of 1-7 the change (if any) they've experienced since beginning treatment in the study (1 = no change or condition has worsened; 7 = a great deal better and a considerable improvement that has made all the difference).
Patient's Global Impression of Change | 20 weeks
  Patient rates on a single item with a scale of 1-7 the change (if any) they've experienced since beginning treatment in the study (1 = no change or condition has worsened; 7 = a great deal better and a considerable improvement that has made all the difference).

OTHER OUTCOMES:
Emotional Approach Coping Scales | Change from baseline to 4 weeks
  Sum of four self-report items assessing whether the subject uses an emotional approach to coping when experiencing stress or difficulties. Items range from 1-4 (1 = I don't use this emotional coping strategy; 4 = I use this emotional coping strategy a lot), yielding a total score between 4 and 16.
Emotional Approach Coping Scales | Change from baseline to 8 weeks
  Sum of four self-report items assessing whether the subject uses an emotional approach to coping when experiencing stress or difficulties. Items range from 1-4 (1 = I don't use this emotional coping strategy; 4 = I use this emotional coping strategy a lot), yielding a total score between 4 and 16.
Emotional Approach Coping Scales | Change from baseline to 20 weeks
  Sum of four self-report items assessing whether the subject uses an emotional approach to coping when experiencing stress or difficulties. Items range from 1-4 (1 = I don't use this emotional coping strategy; 4 = I use this emotional coping strategy a lot), yielding a total score between 4 and 16.
Pain/Brain Attributions Scale | Change from baseline to 4 weeks
  Sum of five self-report items assessing whether the subject beliefs about whether pain is related to stress, brain changes, or emotions. Items range from 0-4 (0 = strongly disagree; 4 = strongly agree) for a total score between 0 and 20.
Pain/Brain Attributions Scale | Change from baseline to 8 weeks
  Sum of five self-report items assessing whether the subject beliefs about whether pain is related to stress, brain changes, or emotions. Items range from 0-4 (0 = strongly disagree; 4 = strongly agree) for a total score between 0 and 20.
Pain/Brain Attributions Scale | Change from baseline to 20 weeks
  Sum of five self-report items assessing whether the subject beliefs about whether pain is related to stress, brain changes, or emotions. Items range from 0-4 (0 = strongly disagree; 4 = strongly agree) for a total score between 0 and 20.
Coping Strategies Questionnaire | Change from baseline to 4 weeks
  Sum of six self-report items assessing the subject's use of coping strategies. Items range 0-6 (0 = never use this strategy; 6 = always use this strategy). Two-item subscales (catastrophizing, increased behavioral activities, cognitive coping) are scored separately, yielding total scores between 0 and 12.
Coping Strategies Questionnaire | Change from baseline to 8 weeks
  Sum of six self-report items assessing the subject's use of coping strategies. Items range 0-6 (0 = never use this strategy; 6 = always use this strategy). Two-item subscales (catastrophizing, increased behavioral activities, cognitive coping) are scored separately, yielding total scores between 0 and 12.
Coping Strategies Questionnaire | Change from baseline to 20 weeks
  Sum of six self-report items assessing the subject's use of coping strategies. Items range 0-6 (0 = never use this strategy; 6 = always use this strategy). Two-item subscales (catastrophizing, increased behavioral activities, cognitive coping) are scored separately, yielding total scores between 0 and 12.
Chronic Pain Acceptance Questionnaire-2 Item | Change from baseline to 4 weeks
  Sum of two self report items assessing the subject's acceptance of chronic pain. Items range from 0-6 (0 = never true; 6 = always true), yielding a total score between 0 and 12.
Chronic Pain Acceptance Questionnaire-2 Item | Change from baseline to 8 weeks
  Sum of two self report items assessing the subject's acceptance of chronic pain. Items range from 0-6 (0 = never true; 6 = always true), yielding a total score between 0 and 12.
Chronic Pain Acceptance Questionnaire-2 Item | Change from baseline to 20 weeks
  Sum of two self report items assessing the subject's acceptance of chronic pain. Items range from 0-6 (0 = never true; 6 = always true), yielding a total score between 0 and 12.
Self-Compassion Scale-Short Form | Change from baseline to 4 weeks
  Sum of twelve self report items assessing the subject's feelings of self-compassion. Items range from 1-5 (1 = almost never; 6 = almost always), yielding a total score between 12 and 60.
Self-Compassion Scale-Short Form | Change from baseline to 8 weeks
  Sum of twelve self report items assessing the subject's feelings of self-compassion. Items range from 1-5 (1 = almost never; 6 = almost always), yielding a total score between 12 and 60.
Self-Compassion Scale-Short Form | Change from baseline to 20 weeks
  Sum of twelve self report items assessing the subject's feelings of self-compassion. Items range from 1-5 (1 = almost never; 6 = almost always), yielding a total score between 12 and 60.
Working Alliance Inventory | Change from baseline to 4 weeks
  Sum of three self-report items assessing the subject's thoughts and feelings on their therapist. Items range 1-7 (1 = never; 4 = sometimes; 7 = always), yielding a total score between 3 and 21.
Working Alliance Inventory | Change from baseline to 8 weeks
  Sum of three self-report items assessing the subject's thoughts and feelings on their therapist. Items range 1-7 (1 = never; 4 = sometimes; 7 = always), yielding a total score between 3 and 21.
Working Alliance Inventory | Change from baseline to 20 weeks
  Sum of three self-report items assessing the subject's thoughts and feelings on their therapist. Items range 1-7 (1 = never; 4 = sometimes; 7 = always), yielding a total score between 3 and 21.
Pain Self-Efficacy Questionnaire-2 item | Change from baseline to 4 weeks
  Sum of two self-report items assessing the subject's confidence in performing activities of daily living despite pain. Items range 0-6 (0 = not at all confident; 6 = completely confident), yielding a total score between 0 and 12.
Pain Self-Efficacy Questionnaire-2 item | Change from baseline to 8 weeks
  Sum of two self-report items assessing the subject's confidence in performing activities of daily living despite pain. Items range 0-6 (0 = not at all confident; 6 = completely confident), yielding a total score between 0 and 12.
Pain Self-Efficacy Questionnaire | Change from baseline to 20 weeks
  Sum of two self-report items assessing the subject's confidence in performing activities of daily living despite pain. Items range 0-6 (0 = not at all confident; 6 = completely confident), yielding a total score between 0 and 12.
Life Events Checklist for DSM-5 | Baseline
  Self report checklist on whether 17 potentially traumatic and life threatening events occurred (yes/no) in the subject's life.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon C Yarns, MD MS BME, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Datasets that meet VA standards for disclosure to the public will be made available within 1 year of publication. Prior to their distribution, a local privacy officer will certify that all datasets contain no PHI. Final datasets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by ORD. Those requesting datasets will be asked to sign a Letter of Agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Datasets that meet VA standards for disclosure to the public will be made available within 1 year of publication. The analytical datasets and statistical code used in publications will be retained for 6 years, in accordance with VA record retention policy.
Access Criteria: Datasets that meet VA standards for disclosure to the public will be made available within 1 year of publication. The analytical datasets and statistical code used in publications will be retained for 6 years, in accordance with VA record retention policy.